CLINICAL TRIAL: NCT04044677
Title: Effect of Combined Virtual Reality Therapy and Transcranial Direct Current Stimulation on Children and Adolescents With Cerebral Palsy.
Brief Title: Virtual Reality Therapy and Transcranial Direct Current Stimulation in Cerebral Palsy.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Talita Dias da Silva, Principal Investigator, University of Sao Paulo
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 99577318.0.0000.5390
Record Dates: First submitted 2019-08-01; First posted 2019-08-05 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: Group 1 will start with ten sessions of tDSC-active combined to VR tasks. After one-month washout, this group will be reallocated to another 10 sessions with tDCS-sham combined to VR tasks. In contrast, Group 2 will do the opposite protocol (participants will start allocated to ten sessions of TDCS-sham and VR tasks, and after one-month washout period will be reallocated to ten sessions of tDCS-active and VR tasks).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The device DS-Stimulator, Neuroconn Mobile tDCS allows the blindness of the researcher and the participant, so the participants, researchers, and outcome assessors will remain blind to group allocation during the study. To ensure proper blinding, participants will receive codes and will be concealed from the allocation process by one different researcher. The researchers responsible for applying the intervention and the outcome assessors will not know the study design, allocation, objectives, and expected outcomes. In addition, for the blinding of the experimenter (responsible for applying the intervention), one assessor (responsible for randomization) will be in charge of giving the active device to the experimenter.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tDSC-active (Experimental): The TDCS-active will be performed over ten consecutive sessions per weekday (i.e. one session daily, no stimulation during the weekend) during the practice of VR games, TDCS-active will be performed with a current of 1 mA and 20 min of duration (20 seconds of ramp-up and ramp-down). The stimulation target will be the M1 area, choosing the more functional side of the participant (C3 or C4).
  This group will perform the tDCS-sham after one-month washout.
  Interventions: Device: tDSC-active
- tDCS-sham (Sham Comparator): The TDCS-sham will be performed over ten consecutive sessions per weekday (i.e. one session daily, no stimulation during the weekend). However, the electrodes will be positioned at the same sites of the tDCS-active and the device will be switched on for 20 seconds (with ramp-up and ramp-down), giving the children the initial sensation of the 1 mA current, but with no stimulation administered during the rest of the time. This sham protocol is already programmed in the device prior to data collection.
  This group will perform the tDCS-active after one-month washout.
  Interventions: Device: tDCS-sham

INTERVENTIONS:
Device: tDSC-active — 10 sessions of active Transcranial Direct Current Stimulation combined to Virtual Reality therapy followed by a one-month washout and 10 sessions of sham Transcranial Direct Current Stimulation
  Arms: tDSC-active
Device: tDCS-sham — 10 sessions of sham Transcranial Direct Current Stimulation combined to Virtual Reality therapy followed by a one-month washout and 10 sessions of active Transcranial Direct Current Stimulation
  Arms: tDCS-sham

SUMMARY:
A double-blinded randomized controlled crossover trial will be conducted, and all participants will undertake non-immersive VR tasks and tDCS-active or tDCS-sham. Group 1 will start with ten sessions of tDSC-active combined to VR tasks. After one-month washout, this group will be reallocated to another 10 sessions with tDCS-sham combined to VR tasks. In contrast, Group 2 will do the opposite protocol (participants will start allocated to ten sessions of TDCS-sham and VR tasks, and after one-month washout period will be reallocated to ten sessions of tDCS-active and VR tasks). All protocol will have the assessment of Autonomic Nervous System, through Heart Rate Variability Analysis.

DETAILED DESCRIPTION:
Study design A double-blinded randomized controlled crossover trial will be conducted, and all participants will undertake non-immersive VR tasks and tDCS-active or tDCS-sham. Group 1 will start with ten sessions of tDSC-active combined to VR tasks. After one-month washout, this group will be reallocated to another 10 sessions with tDCS-sham combined to VR tasks. In contrast, Group 2 will do the opposite protocol (participants will start allocated to ten sessions of TDCS-sham and VR tasks, and after one-month washout period will be reallocated to ten sessions of tDCS-active and VR tasks). The one month washout period has been used in some studies and was shown to be enough to reset the effects of the first ten sessions, considering that the motor effects of the tDCS are sustained from two hours to three months.

Participants and sampling Participants will be recruited through referral by the coordinators of two clinics in Brazil: Intensiva and Therapies. Those interested in participating will undergo a detailed screening against the eligibility criteria for enrollment in the study.

Inclusion criteria Participants will be included if they have the agreement to participate in the research conserve, have a clinical diagnosis of CP done by a neuropediatric clinician with non- progressive etiology (with GMFCS levels I and II and MACS I and II), signing the informed consent form by the parents or guardians.

Exclusion criteria Participants will be excluded if they do not understand the tasks. The understanding of the task will be evaluated through five attempts of each task in VR, because even with low IQ a large part of the adolescents can understand virtual tasks and interact with improved performance.

Dropout criteria Participants will be withdrawn from the study if they are not willing to continue their participation, cannot be present on the day of the experiment or miss two treatment section, and/or change their form of rehabilitation during the study.

Randomization Participants will be randomly allocated to either group 1 (TDCS-active and VR tasks) or group 2 (TDCS-sham and VR tasks) with a 1:1 allocation defined by a computer-generated randomization using the R package (R Foundation for Statistical Computing). Randomization will be under the control of a blinded investigator who will be the only person allowed to manage the electronic security file of the randomization to assign the individuals. The investigator will be blind to the group in which the participant is allocated to.

Blinding The participants, researchers, and outcome assessors will remain blind to group allocation during the study. To ensure proper blinding, participants will receive codes and will be concealed from the allocation process by one different researcher. The researchers responsible for applying the intervention and the outcome assessors will not know the study design, allocation, objectives, and expected outcomes. In addition, for the blinding of the experimenter (responsible for applying the intervention), one assessor (responsible for randomization) will be in charge of giving the active device to the experimenter. The sham device has exactly the same shape of the active. Further details are presented in the "TDCS-sham" section.

Allocation concealment Allocation concealment will successfully be reached since no one involved in this study (i.e. the participants, researchers, and outcome assessors) will be aware of the treatment allocations. Furthermore, investigators will have no control over the order of patients randomized. A blinded investigator will encode the individuals and groups of intervention. To perform the allocation procedure, the encoded groups will be placed inside a closed opaque envelope, which will be labeled with the code for each participant. Envelopes will be opened only during the time of active or sham intervention.

Intervention

All participants will attend the assigned TDCS and VR intervention as follows: there will be twenty sessions over four weeks with TDCS and non-immersive VR tasks, in which ten sessions will be TDCS-active and VR tasks and ten will be TDCS-sham and VR tasks, separated by a one month washout period. The sessions will be administered consecutively and once a day. The researchers will be trained to perform all interventions TDCS-sham, TDCS-active and VR tasks.

Virtual reality intervention. Moreover, after the application of the TDCS-active or Sham, in all sessions will be performed tasks in non-immersive virtual reality environment to stimulate and verify improvement of motor performance. Thus, the "Bridge Games" software tasks will be used. A software developed by the Research and Technological Applications in Rehabilitation (Grupo de Pesquisa e Aplicação Tecnológica em Reabilitação - PATER) group of the School of Arts, Sciences, and Humanities of the University of Sao Paulo (EACH-USP).

Heart Rate Variability HRV analysis will follow the guidelines of the Task Force of the European Society of Cardiology and the North American Society of Pacing and Electrophysiology (TFESC & NASPE, 1996). The strap (for data collection) will be positioned on the participant's chest, and the Polar RS800cx heart rate receiver will be positioned next to it. HRV will be recorded after the initial assessments at rest for 10 minutes, and during virtual reality combined to tDCS training for 20 minutes. For analysis of HRV data at rest 1000 consecutive RR intervals will be used and during the tasks 256 consecutive RR intervals will be used.

HR will be recorded beat by beat throughout the protocol by the Polar RS800CX FC Portable Monitor (Polar Electro, Finland) and RR intervals recorded by the monitor will be transferred to the Polar ProTreiner program (3.0 v., Polar Electro, Finland) , which allows HR visualization and cardiac period extraction in the "txt" file format.

Moderate digital filtering will be performed in the program itself complemented with manual filtering performed in Excel software to eliminate premature ectopic beats and artifacts, and only series with more than 95% sinus beats will be included in the study (Vanderlei et al., 2008).

HRV analysis will be performed using linear (time and frequency domain) and nonlinear methods that will be analyzed using Kubios HRV® software (Kubios HRV v.1.1 for Windows, Biomedical Signal Analysis Group, Department of Applied Physics, University of Kuopio, Finland).

TDCS intervention.

TDCS-active The TDCS-active will be performed over ten consecutive sessions per weekday (i.e. one session daily, no stimulation during the weekend) before the practice of VR games, TDCS-active will be performed with a frequency of 2 Hz and xxxxx pulse trains. The stimulation intensity will be set at 100%..... The stimulation target will be the area associated with the bilateral lower-limb motor area (i.e. vertex, Cz) of the M1.

TDCS-sham The TDCS-sham will be performed over ten consecutive sessions per weekday (i.e. one session daily, no stimulation during the weekend). The TDCS-sham will be used because it ensures the attenuation of stimulous while appearing to be the same device, with good. In addition, the tactile contact of the foam with the skull is maintained.

Procedure During the ETCC protocol, participants will be seated comfortably in a common chair, with their hands arranged over their legs and feet resting on the floor. The demarcation and application of the active TDCS will then be performed in the cortical area corresponding to the primary motor cortex contralateral to the side of the lesion according to EEG System 10-20 (area M1).

Therefore, anodic TDCS with electrodes between 25-35 cm2, intensity of 1 mA, density of up to 0.057 mA / cm2 for a period of 20 minutes will be used. However, for the TDCS-sham (placebo) the same active procedure setting will be used, however, the current will be interrupted after 20 seconds. This configuration will ensure that the electrical stimulus is interrupted before generating considerable stimuli, while the other characteristics of the intervention will be maintained. After each session the participant will be questioned about the presence of adverse effects. The device used will be the DS-Stimulator, from NeuroConn, which allows blindness of the subjects of the research and the experimenters.

After 20 minutes of stimulation, the individuals will perform the training in VR. The training protocol will count on the execution of the following sequence of games: Labyrinth (5 minutes of training with labyrinths of the same dimension, but different ways of solving the task), Memory (5 minutes of training with progressive increase of difficulty according to the number of hits), Fitts (5 minutes) and Interception (5 minutes). The training time will be 20 minutes in total.

Data analysis Considering timing coincident task for the inferential analysis of the initial tasks (transversal) and the longitudinal protocol with ETCC and RV, as dependent variables, the error measures (Constant, Absolute and Variable errors) will be considered (time in milliseconds), if the data meet the assumptions for use of parametric analysis, analysis of variance (ANOVA) will be performed to identify intra and inter-group differences. Differences, if any, will be detected by the post-hoc Tukey-HSD test. If the normality assumptions are not met, non-parametric analyzes will be used to identify and locate the differences: Friedman - post-hoc Wilcoxon as a test (within groups) and Kruskal-Wallis and Mann-Whitney U as a post-hoc test (between groups). For the between groups analysis of HRV indices, it will also be used Multiple Variance Analysis (MANOVA), with repeated measures for within groups analyzes (for evaluations and follow-up) or Mann-Whitney for intergroup analyzes and Friedman for intragroup analyzes. A significance level of 0.05 (5%) will be defined and all intervals constructed throughout the work will be 95% statistical confidence. The statistical program will be SPSS (Statistical Package for Social Sciences), version 26.0.

ELIGIBILITY:
Inclusion Criteria:

* Agreement to participate in the research from their selves and their legal guardians (by signing assent form and consent form);
* Have a clinical diagnosis of CP done by a neuropediatric clinician with non- progressive etiology;
* GMFCS levels I to IV;
* MACS I and IV.

Exclusion Criteria:

* Lack of understanding of the the tasks. The understanding of the task will be evaluated through five attempts of each task in VR, because even with low IQ a large part of the adolescents can understand virtual tasks and interact with improvement of performance;
* Motor difficulties that impede the completing of the virtual tasks;
* Cardiac diseases (because of the HRV assessment).

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2019-01-20 (Actual); Primary Completion 2019-07-20 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Motor skills improvement | 8 weeks.
  The motor skills will be analyzed through the games developed specifically for analysis of motor skills, such as (interception skills, speed, accuracy and reaction time).

SECONDARY OUTCOMES:
Heart Rate Variability | 8 weeks.
  The HRV will be analyzed at rest (20 minutes), during active/sham-tDCS (20 minutes) and during recover from the intervention (10 minutes).

CONTACTS AND LOCATIONS:
Overall Officials: Talita D Silva, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- School of Arts, Sciences and Humanities of the University of Sao Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
We plan to share the study protocol and statistical analysis plan.
Supporting Information: Study Protocol, SAP
Time Frame: Probably from November 1st, forever.
Access Criteria: By accessing the papers published by our group.

REFERENCES:
- [Derived] da Silva TD, Fontes AMGG, de Oliveira-Furlan BS, Roque TT, Lima AII, de Souza BMM, Alberissi CAO, Silveira AC, de Moraes IAP, Collett J, Silva RP, Airoldi MJ, Ribeiro-Papa DC, Dawes H, Monteiro CBM. Effect of Combined Therapy of Virtual Reality and Transcranial Direct Current Stimulation in Children and Adolescents With Cerebral Palsy: A Study Protocol for a Triple-Blinded Randomized Controlled Crossover Trial. Front Neurol. 2020 Sep 2;11:953. doi: 10.3389/fneur.2020.00953. eCollection 2020. PMID 32982950